CLINICAL TRIAL: NCT05919563
Title: Long Term Follow-up of Subjects Who Received GRNOPC1
Brief Title: LTFU Study of Subjects Who Received GRNOPC1
Status: Active, not recruiting | Type: Observational
Sponsor: Lineage Cell Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP35A008
Record Dates: First submitted 2023-05-24; First posted 2023-06-26 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for immune response monitoring and xenotransplantation safety samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects treated with GRNOPC1 in the initial dosing study CP35A007: Subjects treated with GRNOPC1 in the initial dosing study CP35A007 will be followed for 15-year long-term safety monitoring
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Observational study; annual MRI for first 5 years only to monitor changes in the injection site

SUMMARY:
This is a LTFU study for thoracic SCI subjects that were administered GRNOPC1 cells in the main study CP35A007.

DETAILED DESCRIPTION:
Study CP35A008 is a Phase 1, multi-center long term follow-up (LTFU) study for five (5) subjects with complete thoracic SCI that were administered 2 million GRNOPC1 cells in the main study CP35A007. The purpose of this study is to monitor long-term safety in subjects for 15 years post GRNOPC1 administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received administration of GRNOPC1 under clinical study protocol CP35A007.

Exclusion Criteria:

* There are no exclusion criteria for this LTFU study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who received administration of GRNOPC1 under clinical study protocol CP35A007
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-10-06 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Up to 15 years after GRNOPC1 injection
  Information will be collected on all adverse events through Year 5 and on late-occurring adverse events (Years 6-15) related to any changes in neurological condition, a fever of unknown etiology, and the development of neoplasias and/or neurological disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hogge, DVM, MS, PhD, Study Chair — Lineage Cell Therapeutics, Inc.
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Shepherd Center, Atlanta, Georgia
  - Northwestern Medical Group, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McKenna SL, Ehsanian R, Liu CY, Steinberg GK, Jones L, Lebkowski JS, Wirth E, Fessler RG. Ten-year safety of pluripotent stem cell transplantation in acute thoracic spinal cord injury. J Neurosurg Spine. 2022 Apr 1;37(3):321-330. doi: 10.3171/2021.12.SPINE21622. Print 2022 Sep 1. PMID 35364569
- See also: Ten-year safety of pluripotent stem cell transplantation in acute thoracic spinal cord injury — https://pubmed.ncbi.nlm.nih.gov/35364569/